CLINICAL TRIAL: NCT02566876
Title: A Multicentre, Randomised, Double-Blind, Placebo Controlled, Crossover Trial On The Efficacy Of A Mixture Of Three Bifidobacteria In Children With Abdominal Pain-Associated Functional Gastrointestinal Disorders
Brief Title: Bifidobacteria In Children With Abdominal Pain-Associated Functional Gastrointestinal Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Erasmo Miele, Assistant Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02122013
Record Dates: First submitted 2014-02-25; First posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Irritable Bowel Syndrome; Dyspepsia Chronic
Keywords: Children; Abdominal Pain; Functional Dyspepsia; Irritable Bowel Syndrome; Quality of Life
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mixture of three Bifidobacteria (Active Comparator): Patients were administered 1 sachet per day of a mixture of three Bifidobacteria (namely, 3 billions of Bifidobacterium longum BB536®, 1 billion of Bifidobacterium infantis M-63®, and 1 billion of Bifidobacterium breve M-16V®) for six weeks. Subsequently, no preparation was administered for a 2-week-''washout'' period. At each follow-up visit subjects underwent a complete physical examination, data recorded on the daily diaries were collected and compliance to treatment was verified.
  Interventions: Drug: Mixture of three Bifidobacteria
- Placebo (Placebo Comparator): Patients were administered 1 sachet per day of placebo for six weeks. Subsequently, no preparation was administered for a 2-week-''washout'' period. At each follow-up visit subjects underwent a complete physical examination, data recorded on the daily diaries were collected and compliance to treatment was verified.
  Interventions: Drug: Mixture of three Bifidobacteria

INTERVENTIONS:
Drug: Mixture of three Bifidobacteria — This investigation will be a randomized, double-blind, placebo-controlled, cross-over trial. The study will include 70 children with FD or IBS and will be articulated in 16 weeks as follows. Fifty-nine children (median age 11.2 years, range 5.2-17.9) with IBS and FD were randomized to receive either a mixture of three Bifidobacteria or a placebo for 6 weeks. At the end, after a 2-week-''washout'' period, each patient was switched to the other group and followed for 6 further weeks. At baseline and at follow-up, patients and/or their parents completed a dairy for bowel habit and gastrointestinal symptoms, and a quality of life (QoL) questionnaire.
  Other Names: Bifidobacterium infantis M-63® breve M-16V® longum BB536®

SUMMARY:
Abdominal pain (AP)-associated functional gastrointestinal disorders (FGIDs), particularly Irritable Bowel Syndrome (IBS) and Functional Dyspepsia (FD), are common in pediatrics, and no safe and effective treatment is available. Although probiotics have shown promising results in adults, few studies have been published in children. The Bifidobacterium Infantis, Bifidobacterium Breve and Bifidobacterium Longum are the most important beneficial bacteria in children and represent 95% of the total bacterial population in the intestine of breastfed infant.

Objectives: 1) To evaluate the effect of oral administration of a mixture of Bifidobacteria on the improvement of frequency and intensity of AP in children with FD and IBS. 2) To evaluate the effect of oral administration of a mixture of Bifidobacteria on quality of life in children with FD and IBS.

DETAILED DESCRIPTION:
The study was a randomized, double blind, placebo-controlled, crossover trial conducted at two pediatric tertiary care centers in Naples and Foggia. All children aged 8-17 years referred for IBS or FD to the Pediatric Clinics of the two participating centers between January and December 2014 were eligible for the study. IBS and FD were diagnosed using the Rome III criteria for pediatric FGIDs. The main exclusion criterion was the presence of chronic organic gastrointestinal diseases, assessed by full clinical history and examination, and initial laboratory investigation including complete blood cell count, erythrocyte sedimentation rate, C-reactive protein, serum amylase and lipase, tissue transglutaminase antibodies, total serum immunoglubulins A, and fecal calprotectin. Abnormalities in any of these tests resulted in the patient's exclusion from the study. Further exclusion criteria were previous abdominal surgery, diseases affecting bowel motility, or concomitant psychiatric, neurological, metabolic, renal, hepatic, infectious, hematological, cardiovascular or pulmonary disorders. Finally, patients who had been using any commercial preparation of probiotics during the previous 3 months were also excluded.

The study was articulated in 16 weeks. After recruitment, patients entered a 2 week-run-in phase during which evacuative frequency, stool features and gastrointestinal symptoms were recorded on a daily basis using a questionnaire/diary provided at the study entry by the physician. At the end of the baseline period, patients returned to the center where information regarding AP characteristics, bowel habits and associated symptoms were recorded using a previously validated interviewer-administered questionnaire for pediatric FGIDs. The "Functional Disability Inventory" (FDI), a second interviewer-administered validated questionnaire was used to assess physical and psychosocial functions and investigate patients' QoL. The instrument consists of 15 items concerning perceptions of activity limitations during the past 2 weeks; total scores are computed by summing the ratings for each item. Total available score ranges from 0 to 60 and higher scores indicate greater disability. After completing these questionnaires, patients were assigned in a double-blinded fashion to the placebo or intervention group according to a computer-generated randomization allocation table. Participants were randomized to receive either 1 sachet per day of a mixture of three Bifidobacteria (namely, 3 billions of Bifidobacterium longum BB536®, 1 billion of Bifidobacterium infantis M-63®, and 1 billion of Bifidobacterium breve M-16V®), or an identical looking and tasting placebo for six weeks. No further medication other than analgesics was allowed for the whole duration of the study.

After completing the six weeks of treatment, no preparation was administered for a 2-week-''washout'' period. Afterwards, each patient was switched to the other group and treated with placebo or probiotics for a period of six further weeks.

At each follow-up visit subjects underwent a complete physical examination, data recorded on the daily diaries were collected and compliance to treatment was verified. Furthermore, the FGIDs symptoms questionnaire and the FDI were administered by the physician and answers were recorded.

The main outcome parameters considered for the assessment of the efficacy of the administered treatment were abdominal pain and QoL. The investigators considered a decrease in FDI score of at least 75% of the baseline score to define a relevant improvement in QoL. Secondary outcome parameters were changes in bowel habit for IBS patients, and the effect of the tested treatment on nausea for FD subjects.

The investigators involved in the recruitment and follow-up of patients, those coordinating the study and analyzing the data, patients themselves and their caregivers were all unaware of the randomization group at each phase of the study.

The institutional ethical review boards of both participating centers approved the study protocol. Written informed consent was obtained from the parents or legal guardians before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-18years;
* Diagnosis of FD and IBS pain according to the Rome III criteria
* All parents or legal tutors must sign an informed consent document indicating their awareness of the investigational nature of this study.

Exclusion Criteria:

* Taking any other type of probiotic in the 2 months prior to enrollment
* Presence of intestinal motility disorders
* Presence of any other significant medical condition
* Presence of previous abdominal surgery
* Inability or unwillingness to give informed consent

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain Frequency | 16 weeks from the enrollment
  Score ranges from 0 (never) to 5 (every day)

SECONDARY OUTCOMES:
Functional Disability | 16 weeks from the enrollment
  Functional Disability Inventory questionnaire consisting of 15 items concerning perceptions of activity limitations during the previous 2 weeks. Score for each item ranges from 0 (no trouble) to 4 (impossible), for a total score ranging from 0 (no quality of life impairment) to 60 (maximum impairment in quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Giannetti, MD, Principal Investigator — Department of Translational Medical Sciences, Federico II University
Locations (1):
- University of Naples "Federico II" Italy, Naples, Italy

REFERENCES:
- [Derived] Giannetti E, Maglione M, Alessandrella A, Strisciuglio C, De Giovanni D, Campanozzi A, Miele E, Staiano A. A Mixture of 3 Bifidobacteria Decreases Abdominal Pain and Improves the Quality of Life in Children With Irritable Bowel Syndrome: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Crossover Trial. J Clin Gastroenterol. 2017 Jan;51(1):e5-e10. doi: 10.1097/MCG.0000000000000528. PMID 27306945